CLINICAL TRIAL: NCT02822898
Title: Metabolism of Isotonic Versus Hypotonic Maintenance Solutions in Fasting Healthy Adults, a Single-Blind Randomized Crossover Trial
Brief Title: Metabolism of Isotonic Versus Hypotonic Maintenance Solutions in Fasting Healthy Adults
Acronym: MIHMoSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Niels Van Regenmortel, Senior Consultant, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/15/175
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Adult Volunteers
Keywords: Maintenance; Intravenous solutions; Intravenous fluids; Tonicity; Potassium; Sodium; Fluid retention
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotonic Maintenance Fluid (Active Comparator): Isotonic Maintenance Fluid
  Interventions: Drug: NaCl 0.9% in Glucose 5% with 40mEq Potassium
- Hypotonic Maintenance Fluid (Active Comparator): Hypotonic Maintenance Fluid
  Interventions: Drug: Glucion 5%

INTERVENTIONS:
Drug: NaCl 0.9% in Glucose 5% with 40mEq Potassium — NaCl 0.9% in Glucose 5% with 40mEq Potassium, administered at 25 mL/kg IBW/h for 48h
  Arms: Isotonic Maintenance Fluid
Drug: Glucion 5% — Glucion 5% (premixed solution containing 54 mmol/L sodium and 26 mmol/L potassium amongst others), administered at 25 mL/kg IBW/h for 48h
  Arms: Hypotonic Maintenance Fluid

SUMMARY:
The prescription of intravenous maintenance solutions - although widespread - lacks important data on the optimal sodium and potassium content, which has given rise to an important debate in the scientific literature. Our study compares two different infusion fluids in 12 healthy adult volunteers without renal failure in a single-blind randomized crossover design over two 48 hour periods during which subjects are not allowed to eat or drink. Fluid 1 is a premixed solution containing 54 mmol/L of sodium and 26 mmol/L of potassium; fluid 2 is sodium chloride 0.9% in glucose 5% with 40 mmol/L of potassium. Both solutions are administered at 25 mL/kg of ideal body weight, as recommended by current guidelines (NICE 174) and both solutions are widely used in daily clinical practice. The primary hypothesis is that isotonic maintenance solutions lead to more fluid retention than hypotonic fluids. Metabolism of both solutions is assessed by sequential analysis of urine and serum, clinical parameters and bioelectrical impedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, 18-70 years of age
* BMI 17-45 kg/m².
* Creatinine clearance >60 ml/min (according to eGFR CKD-EPI formula).

Exclusion Criteria:

* Acute medical illness within 3 weeks of first study period
* Chronic medication: under diuretic therapy or other chronic medication that interfere with urine output or induce urine retention. All chronic medication should be declared before being enrolled in the study.
* Medical history:

  * cardiac failure,
  * malnourishment,
  * diabetes mellitus,
  * urological disease preventing spontaneous or complete emptying of the bladder,
* any medical or non-medical issue preventing complaint-free fasting for 48 hours (e.g. active peptic ulcer, psychosis, substance abuse…)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Urine Output | 48h
  Urinary output over study period (as AUC).
Body weight | 48h
  Body weight over study period (as AUC), used as a back up parameter for urinary output.

SECONDARY OUTCOMES:
Amount of sodium retention / excretion (excreted sodium / administered sodium) | 48h
  Sodium retention / excretion over study period (mean at 24 and 48h)
Number of episodes of hypokalemia (<3.5 mmol/L), hyponatremia (<135 mmol/L), hypernatremia (>145 mmol/L) | 48h
Change of sodium level from its baseline value. | 48h
  Area under the electrolyte concentration curve (baseline level is reference line)
Change of sodium and potassium level from its baseline value. | 48h
  Area under the electrolyte concentration curve (baseline level is reference line)

OTHER OUTCOMES:
Osmoregulatory Profile 1: urinary volume (mL) | 48h
  Sequential changes in mean urinary volume (per fluid type) at T0-T12-T24-T36-T48.
Osmoregulatory Profile 2: urinary osmolality (mOsm/kg) | 48h
  Sequential changes in mean urinary osmolality (per fluid type). Urinary osmolality is determined on a sample of every individual diuresis. Subjects urinate as the urge rises.
Osmoregulatory Profile 3: serum antidiuretic hormone (ADH) (pg/mL) | 48h
  Sequential changes in mean serum ADH (per fluid type) at T0-T24-T48.
Osmoregulatory Profile 4: thirst score (scale 0-5) | 48h
  Sequential changes in mean thirst score (per fluid type) at T0-T12-T24-T36-T48. The thirst score is a subjective score on a scale of 0-5.
Volume Regulatory Profile 1: urinary sodium (mmol/L) | 48h
  Sequential changes in mean urinary sodium (per fluid type). Urinary sodium is determined on a sample of every individual diuresis. Subjects urinate as the urge rises. Urinary sodium is used to calculate the fractional excretion of sodium.
Volume Regulatory Profile 2: serum aldosterone (ng/dL) | 48h
  Sequential changes in mean serum aldosterone (per fluid type) at T0-T24-T48.
Volume Regulatory Profile 3: urinary potassium (mmol/L) | 48h
  Sequential changes in mean urinary potassium (per fluid type). Urinary potassium is determined on a sample of every individual diuresis. Subjects urinate as the urge rises.
Acid-Base Profile 1: serum chloride (mmol/L) | 48h
  Sequential changes in mean serum chloride (per fluid type) at T0-T12-T24-T36-T48.
Acid-Base Profile 2: serum apparent strong ion difference (mEq/L) | 48h
  Sequential changes in mean serum apparent strong ion difference (per fluid type) at T0-T12-T24-T36-T48.
Acid-Base Profile 3: urinary anion gap (mmol/L) | 48h
  Sequential changes in mean urinary anion gap (per fluid type). Urinary potassium is determined on a sample of every individual diuresis. Subjects urinate as the urge rises.
Other Electrolytes Profile 1: Serum phosphate (mmol/L) | 48h
  Sequential changes in mean serum phosphate (per fluid type) at T0-T24-T48.
Other Electrolytes Profile 2: Red blood cell magnesium (mmol/L) | 48h
  Sequential changes in mean red blood cell magnesium (per fluid type) at T0-T24-T48.
Cortisol (µg/dL) | 48h
  Serum cortisol as a measure of stress due to fasting.
Bioelectrical impedance analysis 1: Total body water | 48h
  Sequential changes in mean total body water (per fluid type) at T0-T24-T48.
Bioelectrical impedance analysis : Extracellular volume | 48h
  Sequential changes in mean extracellular volume (per fluid type) at T0-T24-T48.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Van Regenmortel, M.D., Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital, Antwerp, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lobo DN, Bostock KA, Neal KR, Perkins AC, Rowlands BJ, Allison SP. Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet. 2002 May 25;359(9320):1812-8. doi: 10.1016/S0140-6736(02)08711-1. PMID 12044376
- [Background] Moritz ML, Ayus JC. Maintenance Intravenous Fluids in Acutely Ill Patients. N Engl J Med. 2015 Oct;373(14):1350-60. doi: 10.1056/NEJMra1412877. No abstract available. PMID 26422725
- [Derived] Van Regenmortel N, De Weerdt T, Van Craenenbroeck AH, Roelant E, Verbrugghe W, Dams K, Malbrain MLNG, Van den Wyngaert T, Jorens PG. Effect of isotonic versus hypotonic maintenance fluid therapy on urine output, fluid balance, and electrolyte homeostasis: a crossover study in fasting adult volunteers. Br J Anaesth. 2017 Jun 1;118(6):892-900. doi: 10.1093/bja/aex118. PMID 28520883
- See also: NICE guideline on Intravenous Fluid Therapy in Adults in Hospital — http://guidance.nice.org.uk/CG174
- See also: GIFTASUP guidelines — http://www.bapen.org.uk/pdfs/bapen_pubs/giftasup.pdf